CLINICAL TRIAL: NCT04617600
Title: Survival Rate After TheraCal PT Pulpotomy Versus MTA Pulpotomy in Children With Vital Primary Molars: A Randomized Controlled Pilot Trial.
Brief Title: Survival Rate After TheraCal PT Pulpotomy Versus MTA Pulpotomy in Children With Vital Primary Molars.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Reem Mohamed Gaber, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14422019496708
Record Dates: First submitted 2020-10-22; First posted 2020-11-05 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: Reversible Pulpitis
MeSH Terms: interventions — Pemetrexed; mineral trioxide aggregate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mineral trioxide aggregate (MTA) (Active Comparator): Survival rate of cariously exposed vital primary molars using MTA+ Curamed (UI, Kwiatkowskiego 1, 37-450 Staleya Wola, Polka)
  Interventions: Drug: MTA
- TheraCal PT (Experimental): Survival rate of cariously exposed vital primary molars using TheraCal PT (BISCO Dental Products, Schamberg IL, U.S.A.)
  Interventions: Drug: TheraCal PT

INTERVENTIONS:
Drug: MTA — Survival rate using MTA in cariously exposed vital primary molars
  Other Names: Mineral trioxide aggregate
  Arms: Mineral trioxide aggregate (MTA)
Drug: TheraCal PT — Survival rate using TheraCal PT in cariously exposed vital primary molars
  Other Names: TheraCal PT®
  Arms: TheraCal PT

SUMMARY:
The aim of the study is to assess the effect of TheraCal PT pulpotomy versus MTA pulpotomy on the survival rate of cariously exposed vital primary molars.

DETAILED DESCRIPTION:
for both interventions ,

1. Informed consent from participating parents.
2. Baseline records photographs, percussion test, periapical radiograph and personal data collection.
3. Allocation (concealed by withdrawing a sealed opaque envelope containing eight times folded paper containing the type of dressing material that will be used then writing patient name and I.D. on it and will be opened after performing the access cavity).
4. Diagnostic chart with personal, medical and dental history will be filled.
5. Clinical examination will be performed to assess the clinical inclusion criteria. (Pulpal and periapical diagnosis is established after clinical examination).
6. Preoperative and Postoperative photographs will be taken.
7. The radiographic examination will be performed by taking periapical x-ray using (parallel technique) through machine to assess the inclusion criteria. The preoperative radiograph will serve as a reference for the follow-up radiographs. Standardization of the technique to avoid any distortion in the vertical dimension and to provide reproducible images using x-ray holding device.
8. Preoperative and postoperative radiograph will be taken by parallel technique using extension cone paralleling (XCP) film holder.
9. Administration of inferior alveolar nerve block (Septodont, Scandonest® 2% L Mepivacaine hydrochloride (HCl). 2% and Levonordefrin 1:20,000 Injection, U.S.P.) at the side of the affected tooth.
10. Application of rubber dam for isolation, then a standardized pulpotomy procedure will be performed using a large sterile round end bur in a high-speed handpiece with copious irrigation, a sharp spoon excavator will remove pulpal tissues to the orifice level. Hemostasis will be achieved by the application of a wet cotton pellet.

Children will then be allocated into either one of the groups alternatively depending on the pulpotomy medicament used as follows:

* Group I (Experimental group) TheraCal PT pulpotomy.
* Group II (Control group) MTA pulpotomy.

Group I (Experimental group) TheraCal PT:

1. After complete hemostasis, TheraCal PT (BISCO Dental Products, Schamberg illinois (IL), U.S.A.) will be applied according to the manufacturer's instructions and gently placed over the pulp stumps to a thickness of 2mm then the rest of the pulp chamber will be filled with glass ionomer cement.
2. Tooth will then be restored with stainless steel crown.

Group II (Control group) MTA pulpotomy:

1. After complete hemostasis, MTA+ Curamed (ul. Kwiatkowskiego 1, 37-450 stylosa Wola, Polka) will be manipulated in the ratio of 3:1 (powder: liquid) to obtain a putty mix. This mix will be placed over the radicular pulp with the help of a suitable sterile amalgam carrier. Gentle condensation of the mix will be done in the pulp chamber with a moistened cotton pellet, followed by application of glass ionomer cement.
2. Tooth will then be restored with stainless steel crown.

ELIGIBILITY:
Inclusion Criteria:

* Aged 4 to 7 years , in good general health and mentally free.
* The parents provided written informed consent.
* Cariously exposed primary molars with reversible pulpitis.
* Teeth should be vital.
* Restorable teeth.
* Hemostasis achieved after complete pulpotomy

Exclusion Criteria:

* With systemic disease.
* Physical or mental disability.
* Unable to attend follow-up visits.
* Refusal of participation.
* Previously accessed teeth.
* History of spontaneous or prolonged pain.
* Swelling, tenderness to percussion or palpation, or pathological mobility.
* Pre-operative radiographic pathology such as resorption(internal or external),per-radicular or furcation radiolucency.
* Haemorrhage control is unachievable after pulpotomy.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Survival rate (Absence of spontaneous pain) | "3 months"
  Binary outcome measured with direct questioning to the patient
Survival rate (Absence of spontaneous pain) | "6 months"
  Binary outcome measured with direct questioning to the patient
Survival rate (Absence of swelling) | "3 months"
  Binary outcome measured visually by intraoral/extraoral examination
Survival rate (Absence of swelling) | "6 months"
  Binary outcome measured visually by intraoral/extraoral examination

SECONDARY OUTCOMES:
Absence of periapical radiolucency or absence of internal/external root resorption | "6 months"
  Binary outcome detected with periapical x-ray by parallel technique using XCP film holder (Super Bite, Hawe Neos DentalSA, Switzerland).
Time lapse till final restoration performed. | "During procedure".
  Continuous outcome measured with a Stopwatch in minutes.

IPD SHARING:
Plan to Share IPD: No